CLINICAL TRIAL: NCT02785562
Title: Epidemiologic Multicenter Prospective Study in Advanced NSCLC Patients With PDL1 Expression : Evaluation of Clinical and Pathological Characteristics of PDL1 High Expression Patients Compared to Patients With a Weak or no Expression of PDL1.
Brief Title: Epidemiologic Multicenter Prospective Study in Advanced NSCLC (Non Small Cell Lung Cancer) Patients With PDL1 (Protein Death Ligand 1) Expression.
Acronym: EXPLORE-PDL1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GFPC 06-2015
Record Dates: First submitted 2016-03-01; First posted 2016-05-30 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer
Keywords: PDL1 expression : Protein Death Ligand 1 expression .
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assessment of PDL1 expression (Other): Other : assess clinical and pathological characteristics of PDL1 expression in Non Small Cell Lung Cancer patients.
  Interventions: Other: Assessment of PDL1 expression

INTERVENTIONS:
Other: Assessment of PDL1 expression — Intervention : 2 biopsy slides will be analyzed in central laboratory.

SUMMARY:
Epidemiologic multicenter prospective study in advanced NSCLC patients with PDL1 expression : evaluation of clinical and pathological characteristics of PDL1 high expression patients compared to patients with a weak or no expression of PDL1.

DETAILED DESCRIPTION:
Few data are published on the clinical and pathological characteristics of advanced NSCLC with high PDL1 expression compare to weak and no expression populations.

There is not for the moment a standard test to determine a relevant target population. Preliminary data showed that around 25% of the NSCLC population may have a high PDL1 expression and may have a greater benefit of anti PDL1 therapy. But in fact limited data have been published in European populations on the clinical and pathological characteristics (high PDL1 expression) compared to the weak expression and no expression populations. More over the prognosis rule of a high PDL1 expression in NSCLC is not definitive, with some studies indicating it is a positive prognostic factor while other studies showing that it is a negative prognostic factor.

To understand if there are differences in terms of prognostic between advanced NSCLC with high and low/no expression of PDL1 is a major challenge for the future management strategy of these patients. The results of this study should helps to elaborate new guidelines for this population. Therefore is also important to had data's on the natural course of the disease in these population for building cost effectiveness models of new immune therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more

  * With locally advanced stage (IIIb) to stage IV NSCLC - Non Small Cell Lung Cancer -
  * Histological diagnostic :
* No known Epidermal Growth Factor Receptor (EGFR) or Anaplastic Lymphoma Kinase (ALK) / Reactive Oxygen Species (ROS) translocation
* At least 2 slides of tumoral sample available

  * No previous chemotherapy treatment. Neo or adjuvant therapy is allowed if done at least one year before inclusion
  * Performance Status ( PS) 0/1

Planned to receive a platin based standard treatment (cisplatin or carboplatin with bevacizumab (restricted to no squamous) pemetrexed(restricted to no squamous) , gemcitabine, vinorelbine, docetaxel or taxol, on first line setting, in standard dose

• A RECIST - Response Evaluation Criteria In Solid Tumor - target lesion

Exclusion Criteria:

* Age fewer than 18
* Pregnancy
* Known immune deficit
* PS > 1
* Inclusion in a clinical therapeutic trial in first line
* Patient treated with Protein D1/Protein Death Ligang1 (PD1/PDL1) therapy on first line setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-06 (Actual)

PRIMARY OUTCOMES:
description of the PDL1 expression groups as follows : PDL1 negative, PDL1 positive, PDL1 weak, PDL1 strongly positive. | 24 Months
  Descriptive and comparative analyses of different sub-populations will be performed with qualitative and quantitative variables. Quantitative variables will be described using the following descriptive statistics: sample size, number of missing values, mean, standard deviation, median, minimum and maximum.
  Qualitative variables will be described using the following descriptive statistics: sample size, number of missing values and percentage of each modality calculated from the responses expressed.
  The bivariate statistical analyses performed will be subjected to statistical tests, based on the nature of the variables analyzed.
Clinical characteristics of PDL1 high expression patients compared to patients with a weak or no expression of PDL1. | 24 Months
  Descriptive and comparative analyses of different sub-populations will be performed with qualitative and quantitative variables. Quantitative variables will be described using the following descriptive statistics: sample size, number of missing values, mean, standard deviation, median, minimum and maximum.
  Qualitative variables will be described using the following descriptive statistics: sample size, number of missing values and percentage of each modality calculated from the responses expressed.
  The bivariate statistical analyses performed will be subjected to statistical tests, based on the nature of the variables analyzed.
Pathological characteristics of PDL1 high expression patients compared to patients with a weak or no expression of PDL1. | 24 Months
  Descriptive and comparative analyses of different sub-populations will be performed with qualitative and quantitative variables. Quantitative variables will be described using the following descriptive statistics: sample size, number of missing values, mean, standard deviation, median, minimum and maximum.
  Qualitative variables will be described using the following descriptive statistics: sample size, number of missing values and percentage of each modality calculated from the responses expressed.
  The bivariate statistical analyses performed will be subjected to statistical tests, based on the nature of the variables analyzed.

SECONDARY OUTCOMES:
Clinical analysis of the patients' outcome : measure of Overall Survival (OS). | 24 Months
  Descriptive and comparative analyses of different sub-populations will be performed with qualitative and quantitative variables. Quantitative variables will be described using the following descriptive statistics: sample size, number of missing values, mean, standard deviation, median, minimum and maximum.
  Qualitative variables will be described using the following descriptive statistics: sample size, number of missing values and percentage of each modality calculated from the responses expressed.
  The bivariate statistical analyses performed will be subjected to statistical tests, based on the nature of the variables analyzed.
Immune characteristics of high PDL1 expression, concordance between PDL1 expression and description of immune environment measured through density of the intra tumoral Cluster of differentiation 8+ lymphocyte T cell (CD8+ Tcells/mDC). | 24 Months
  The density of tumoral T cells will be described in the overall population and each subgroup through descriptive statistics. The Chi2 test will be used to assess the significance of the difference between the different subgroups.
Quality of life of the patients measured at each cycle of therapy thanks to EuroQol Group 5-Dimension Self-Report Questionnaire score (EQ5D questionnaire). | 24 Months
  A descriptive analysis of the answers to the EQ5D will be performed. Evolution of the EQ5D profile will be evaluated. Exploratory analyzes of various risk factors of impaired quality of life will be realized. The proportion of patients reporting "no", "some", or "extreme" EQ5D health state profiles at pre-specified time points will be described.
Measure of the Health Care Resource Use (HCRU) associated to the management of the patients thanks to EQ5D (EuroQol Group 5-Dimension Self-ReportQuestionnaire score) questionnaire. | 24 Months
  Health Care Resource Use consumption will be measured associated to EQ5D questionnaire answers.

CONTACTS AND LOCATIONS:
Overall Officials: Christos CHOUAID, Professor, Principal Investigator — FCPC Vice President
Locations (13):
- France (13):
  - Centre Hospitalier D Argenteuil, Argenteuil, VAL D'oise
  - Site 12, Aix-en-Provence
  - Centre Hospitalier Universitaire, Angers
  - Site 22, Beauvais
  - Centre Hospitalier du Morvan, Brest
  - Site 48, Clermont-Ferrand
  - Site 33, Créteil
  - Site 04, Gap
  - Centre Hospitalier Les Oudairies, La Roche-sur-Yon
  - Centre Hospitalier Universitaire DUPUYTREN, Limoges
  - Site 19, Périgueux
  - Site 18, Rouen
  - Site 11, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fong L, Small EJ. Anti-cytotoxic T-lymphocyte antigen-4 antibody: the first in an emerging class of immunomodulatory antibodies for cancer treatment. J Clin Oncol. 2008 Nov 10;26(32):5275-83. doi: 10.1200/JCO.2008.17.8954. Epub 2008 Oct 6. PMID 18838703
- [Result] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- Available data/document: Study Protocol — http://www.g-f-p-c.org — The login can be obtained directly on gfpc site.